CLINICAL TRIAL: NCT01616901
Title: Wean Obese Study : Determination of the Optimal Spontaneous Breathing Trial for Obese Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8923
Record Dates: First submitted 2012-06-04; First posted 2012-06-12 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2012-06

CONDITIONS: Obesity; Respiratory Failure; PSV 7cmH2O PEEP 7cmH2O; PSV 7 cmH2O PEEP 0 cmH20; CPAP 7 cmH2O; PSV 0 cmH20 PEEP 0 cmH2O; T-Tube; Post-extubation in Spontaneous Breathing and/or in NIV
Keywords: Obese; Intensive Care; Respiratory weaning; Spontaneous Breathing trial; Work of breathing
MeSH Terms: conditions — Obesity; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Spontaneous breathing trial (Experimental)
  Interventions: Procedure: Spontaneous breathing trial

INTERVENTIONS:
Procedure: Spontaneous breathing trial — 5 spontaneous breathing trial will be tested by the patients in the same order :
  * 7 cm H2O continuous positive airway pressure
  * T piece
  * 7 cmH2O of pressure support
  * 0 cmH20 of pressure support
  * 7 cm H2O pressure support ventilation with 7 cmH20 of end expiratory pressure.

SUMMARY:
The decision to extubate a patient after acute respiratory failure is based on clinical observation and measurement of pulmonary mechanics. Current extubation criteria(tidal volume, respiratory frequency...) lack of specificity. The best way to evaluate and predict patients breathing abilities after extubation is to challenge him to a spontaneous breathing trial (SBT) with endotracheal tube in place immediately before extubation to predict the patient's ability to breathe spontaneously after extubation. The intention is to approximate, while the patient is still intubated, the work of breathing that will be required of the patient after extubation. Different approaches of ventilatory settings are currently used for the preextubation SBT, whether pressure support ventilation (PSV), continuous positive airway pressure (CPAP), or spontaneous ventilation through an endotracheal tube (T piece), all supported by literature with different benefits. To the investigators knowledge, few studies define which mode of ventilation most closely approximates the work of breathing during spontaneous respiration after extubation, and none have studied a specific population of obese patient in respiratory weaning. The main objective of the investigators study is to determine, between five different SBT, which one is the best to approximate the work of breathing of obese patient after extubation.

DETAILED DESCRIPTION:
Patients : 20 obese patients (defined by BMI over 30 kg/m2) ongoing for spontaneous breathing trial and clinically ready for immediate extubation will be enrolled after obtaining their consents. Material : An oeso-gastric double balloon catheter will be inserted in order to record oesophageal and gastric pressure and to calculate Work of Breathing and Pressure Time Product. Pulmonary Volumes will be recorded by a pneumotachograph. Functional Residual Capacity will be recorded thanks to the azote double dilution technique used by the Engström respiratory care station.Study Protocol : When physicians in charge of the patient decided that the patient is ready to be weaned and to have a SBT before extubation, the patient will be included in the study. Before extubation, patients will be placed under 5 different spontaneous breathing trials conditions in the same order : 7 cm H2O continuous positive airway pressure, T piece,7 cmH2O of pressure support, 0 cmH20 of pressure support and 7 cm H2O pressure support ventilation with 7 cmH20 of end expiratory pressure. Each trial will be performed fo 20 min. Between 2 spontaneous breathing trials, and before extubation, patient will receive a 10 minutes period of recovery to their respiratory baseline, defined by the respiratory settings before the spontaneous breathing trials.The last step, after extubation, will consist in recording the data after 15 minutes, when patient's breathing pattern appears calm.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 kg/m2
* Weaning procedure achieved, ongoing for extubation

Exclusion Criteria:

* Contra indication for nasogastric catheter placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Work of breathing | Duration of hospital stay: one day
  Based upon the Campbell diagram, WOB will be calculated by integrating oesophageal pressure to tidal volume in time.

SECONDARY OUTCOMES:
Functional Residual Capacity | Duration of hospital stay: one day
  Lung recruitement will be evaluated by a bed side technique of FRC mesurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology & Critical Care, St Eloi University Hospital, Montpellier, France

REFERENCES:
- [Derived] Mahul M, Jung B, Galia F, Molinari N, de Jong A, Coisel Y, Vaschetto R, Matecki S, Chanques G, Brochard L, Jaber S. Spontaneous breathing trial and post-extubation work of breathing in morbidly obese critically ill patients. Crit Care. 2016 Oct 27;20(1):346. doi: 10.1186/s13054-016-1457-4. PMID 27784322